CLINICAL TRIAL: NCT02650882
Title: Effect of Inspiratory Muscle Training on the Performance of Handball Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Charlini Simoni Hartz, Principal Investigator, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 62/13
Record Dates: First submitted 2015-11-10; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Athletic Performance
Keywords: Respiratory muscles; athletic performance; handball

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Placebo group (PG) Nine athletes who maintained their regular sporting activities and were submitted to the IMT program for 12 weeks with a fixed load at 15% MIP, placebo protocol.
  Interventions: Procedure: Device POWERbreathe
- Experimental (Experimental): Experimental group (EG) Ten athletes who maintained their regular sporting activities and were submitted to the IMT program for 12 weeks with a progressive load at 60%, 70% and 80 % of MIP.
  Interventions: Procedure: Device POWERbreathe

INTERVENTIONS:
Procedure: Device POWERbreathe

SUMMARY:
This study investigated the effects of an inspiratory muscle training (IMT) program on the respiratory muscle strength and resistance and the aerobic physical performance (PP) of handball athletes. Nineteen male athletes took part in the study, allocated at random into the experimental group (EG, n=10) and the placebo group (PG, n=9), aged 19±1 and 22±5 years old, respectively. The respiratory muscle strength (RMS) was evaluated by measuring the maximum inspiratory and expiratory pressures (MIP and MEP, respectively), the muscular respiratory resistance was evaluated by maximum voluntary ventilation (MVV) and the aerobic PP by applying the cardiopulmonary exercise test. Subsequently the volunteers were submitted to an IMT protocol 5 times a week for 12 weeks.

DETAILED DESCRIPTION:
The study was designed to evaluate the effects of a 12-week IMT program on the respiratory muscle strength and aerobic physical performance of handball players. Nineteen male athletes took part in the study, divided into the experimental group (EG), which took part in the evaluations, maintained their regular sporting activities and carried out the IMT (n=10), and the placebo group (PG), which took part in the evaluations, maintained their regular sporting activities and carried out an IMT with a load considered to be placebo (n=09), Experimental procedures were carried out by trained researchers and a qualified team. The evaluations and IMT were carried out during the competitive season, the training frequency being based on the competition program, following the traditional annual model.

The athletes were submitted to an initial evaluation composed of measuring the respiratory muscle strength (RMS) using a manovacuometer, and an evaluation of the aerobic physical performance carried out using the cardiopulmonary exercise test (CPET).

The athletes were reevaluated after 12 weeks for subsequent analysis and comparison with the initial values.

All the subjects were previously informed about the experimental procedures, and signed a free and clarified term of consent. The project was approved by the Ethics in Research Committee of the Institution with the number 62/13.

ELIGIBILITY:
GENDER: Male

AGE LIMITS:

Minimum age: 18 years Maximum age:30 years Accepts Healthy Volunteers? YES

Eligibility Criteria

Inclusion criteria:

* male gender
* competition level athlete for at least one year
* regularly takes part in the training sessions

Exclusion criteria:

* smoke
* shows signs of respiratory and/or cardiovascular diseases
* use supplements and/or medication that influences physical performance

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effect of inspiratory muscle training on the respiratory muscle strength performed using a manometer and measured with cmH20 | Finalized study (24 weeks)
  The evaluation of respiratory muscle strength (RMS) was performed using a manometer and measured with cmH20
Effect of inspiratory muscle training on the muscular respiratory resistance evaluated by maximum voluntary ventilation (MVV) carried out with a spirometer | Finalized study (24 weeks)
  The muscular respiratory resistance was evaluated by maximum voluntary ventilation (MVV) carried out with a spirometer
Effect of inspiratory muscle training on the aerobic physical performance (PP) using cardiopulmonary test (CPT), and measured by VO2max | Finalized study (24 weeks)
  The evaluation of aerobic performance was carried out using cardiopulmonary test (CPT), and measured by VO2max